CLINICAL TRIAL: NCT04253431
Title: A Single-blind, Randomized, Single-centre Study to Investigate the Characteristics of Different Personal Lancets on Blood Volume and Perceived Pain in Patients With Diabetes Mellitus
Brief Title: The Characteristics of Different Personal Lancets on Blood Volume and Perceived Pain in Patients With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HTL-Strefa S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: mp08.13
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: lancing device; lancet; fingerprick; capillary blood; self-monitoring of blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- L01 (Experimental): Finger pricking using lancing device with personal lancets
  Interventions: Device: Droplet lancing device (HTL-Strefa S.A.); Device: Ultra-Fine 33G lancets (BD)
- L02 (Experimental): Finger pricking using lancing device with personal lancets
  Interventions: Device: Microlet 2 lancing device (Bayer); Device: Droplet 33G lancets (HTL-Strefa S.A.)
- L03 (Experimental): Finger pricking using lancing device with personal lancets
  Interventions: Device: OneTouch Delicia lancing device (LifeScan); Device: OneTouch Delicia Extra Fine 33G lancets (LifeScan)
- L04 (Experimental): Finger pricking using lancing device with personal lancets
  Interventions: Device: Droplet lancing device (HTL-Strefa S.A.); Device: HaemoFine 33G lancets (HTL-Strefa S.A.)
- L05 (Experimental): Finger pricking using lancing device with personal lancets
  Interventions: Device: ReliOn lancing device (ReliOn); Device: ReliOn Ultra-Thin Plus 33G lancets (ReliOn)
- L06 (Experimental): Finger pricking using lancing device with personal lancets
  Interventions: Device: Accu-Chek Softclix lancing device (Roche); Device: Softclix 28 G lancets (Roche)
- L07 (Experimental): Finger pricking using lancing device with personal lancets
  Interventions: Device: Microlet 2 lancing device (Bayer); Device: Microlet 28G lancets (Bayer)
- L08 (Experimental): Finger pricking using lancing device with personal lancets
  Interventions: Device: Droplet lancing device (HTL-Strefa S.A.); Device: Droplet 33G lancets (HTL-Strefa S.A.)
- L09 (Experimental): Finger pricking using lancing device with personal lancets
  Interventions: Device: BGStar lancing device (Sanofi Aventis); Device: BGStar Ultra-Thin 33G lancets (Sanofi Aventis)
- L10 (Experimental): Finger pricking using lancing device with personal lancets
  Interventions: Device: HaemoFine 33G lancets (HTL-Strefa S.A.); Device: GlucoJect Dual S lancing device (Menarini)

INTERVENTIONS:
Device: Droplet lancing device (HTL-Strefa S.A.)
  Arms: L01; L04; L08
Device: Microlet 2 lancing device (Bayer)
  Arms: L02; L07
Device: OneTouch Delicia lancing device (LifeScan)
  Arms: L03
Device: ReliOn lancing device (ReliOn)
  Arms: L05
Device: Accu-Chek Softclix lancing device (Roche)
  Arms: L06
Device: BGStar lancing device (Sanofi Aventis)
  Arms: L09
Device: Ultra-Fine 33G lancets (BD)
  Arms: L01
Device: Droplet 33G lancets (HTL-Strefa S.A.)
  Arms: L02; L08
Device: OneTouch Delicia Extra Fine 33G lancets (LifeScan)
  Arms: L03
Device: HaemoFine 33G lancets (HTL-Strefa S.A.)
  Arms: L04; L10
Device: Softclix 28 G lancets (Roche)
  Arms: L06
Device: ReliOn Ultra-Thin Plus 33G lancets (ReliOn)
  Arms: L05
Device: GlucoJect Dual S lancing device (Menarini)
  Arms: L10
Device: Microlet 28G lancets (Bayer)
  Arms: L07
Device: BGStar Ultra-Thin 33G lancets (Sanofi Aventis)
  Arms: L09

SUMMARY:
A randomized single-blind study with the use of different lancing devices equipped with personal lancets to determine and to compare the amount of capillary blood volume and perceived pain after a single lancing of the fingertip.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the informed consent.
* Must currently be diagnosed with either Type I or Type II diabetes mellitus.
* Otherwise in good physical and mental health.
* Must currently be performing self-monitoring of blood glucose (self reported).
* Must be between 18-75 years of age (inclusive).
* Ability to read and follow study instructions.

Exclusion Criteria:

* Pregnancy (self reported).
* Severe poor blood circulation in the fingers.
* Any skin condition on his or her fingers that prevents blood sampling.
* History of a bleeding disorder.
* Neuropathy or other condition affecting sensation in the hands.
* Self-reported blood borne infection (e.g., HIV, hepatitis B or C, syphilis, malaria, babesiosis, brucellosis, leptospirosis, arboviral infections, relapsing fever, T lymphotropic virus Type 1, Creutzfeldt-Jakob disease).
* Currently participating in another study.
* History of drug or alcohol abuse within the 12 months prior to screening or evidence of such abuse.
* Donation or loss of 400 mL or more of blood within 4 weeks prior to the start of the study.
* Any prescription or OTC medication within two days of starting the study which might affect pain perception (for example, ibuprofen or paracetamol).
* Alcohol 48 hours before study start.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Volume (uL) of blood in the capillary tube | The blood from the puncture site was collected to the capillaries for 30 seconds, and afterwards amount of the blood was measured using a calibrated ruler
  Examination of the volume of blood obtained after puncturing a fingertip with the use of different lancing devices set to maximum puncture depth, with the use of various-sized personal lancets (28G and 33G).

SECONDARY OUTCOMES:
The intensity of pain perceived by the patient assessed with the use of the VAS (Visual Analog Scale). | 3 minutes (+/- 1 minute) after lancing
  Examination of the intensity of pain perceived when puncturing a fingertip with the use of different lancing devices set to maximum puncture depth, with the use of various-sized personal lancets (28G and 33G).